CLINICAL TRIAL: NCT01895374
Title: A Comparison of the Effects of Bovine Freeze-dried Amniotic Membrane and Hydrocolloid on Epithelialization After Laser Treatments
Brief Title: Clinical Efficacy of Bovine Freeze-dried Amniotic Membrane on Wound Healing in Laser Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0320
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Biological Dressings
Keywords: Laser therapy; Biological dressing; Amniotic membrane; Hydrocolloid bandages; wound healing
MeSH Terms: interventions — Laser Therapy; Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- amniotic membrane dressing (Experimental): We compare the efficacy of amniotic membrane and hydrocolloid in same subjects to avoid confounders.
  Interventions: Procedure: laser treatments; Other: amniotic membrane application
- Hydrocolloid dressing (Active Comparator): Same subjects received amniotic membrane and hydrocolloid dressing at the same time in different wound.
  Interventions: Procedure: laser treatments; Device: hydrocolloid application

INTERVENTIONS:
Procedure: laser treatments
  Other Names: Laser ablation of the skin lesions
Other: amniotic membrane application
  Other Names: dressing with amniotic membrane
  Arms: amniotic membrane dressing
Device: hydrocolloid application
  Other Names: dressing with hydrocolloid as a comparator
  Arms: Hydrocolloid dressing

SUMMARY:
Bovine amniotic membrane may show better efficacy than hydrocolloid dressing.

DETAILED DESCRIPTION:
Bovine amniotic membrane as a biological dressing can be applicable to wound after laser treatments. Comparing with hydrocolloid dressing material, which is the most widely used after laser treatment now, amniotic membrane will show better efficacy. Thus, with amniotic membrane, epithelization time will shorten and redness which is usually left after laser will disappear quickly.

ELIGIBILITY:
Inclusion Criteria:

* Skin lesions treatable by ablative lasers
* More than two skin lesions of similar size at the same area
* Available during the study period (2 weeks)

Exclusion Criteria:

* Taking steroid or nonsteroidal antiinflammatory drug, isotretinoin
* underlying diabetes mellitus, keloid or any malignancy

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2012-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Epithelization time | 2 weeks
  time to complete epithelization after wounding

SECONDARY OUTCOMES:
Epithelization Scale | 2 weeks
  Assessment of redness, oozing, swelling
Photometric measurements | 2 weeks
  spectrophotometer and colorimeter
Vancouver scar scale | 2 weeks
  Vancouver scar scale
Assessment by subjects | 2 weeks
  pain, itching, inconvenience
measurements of adverse effects | 2 weeks
  assessments of adverse effects by investigator
histopathologic analysis | 2 weeks
  changes of the tissue with time

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hun Suh, PhD, Study Chair — Department of Dermatology, Seoul National University College of Medicine; Seonguk Min, Msc, Principal Investigator — Department of Dermatology, Seoul National University College of Medicine
Locations (1):
- Department of Dermatology, Seoul National University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Singh R, Chacharkar MP. Dried gamma-irradiated amniotic membrane as dressing in burn wound care. J Tissue Viability. 2011 May;20(2):49-54. doi: 10.1016/j.jtv.2010.06.001. Epub 2010 Jul 8. PMID 20619656